CLINICAL TRIAL: NCT02011594
Title: Phase II Study of Maintenance Treatment of Nimotuzumab Versus No Maintenance for Advanced Esophageal Carcinoma
Brief Title: Phase II Study of Maintenance Treatment of Nimotuzumab for Advanced Esophageal Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There was no participants enrolled in this clinical trial.
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1407
Record Dates: First submitted 2013-12-07; First posted 2013-12-13 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Stage IV Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Nimotuzumab
  Interventions: Drug: Nimotuzumab
- Arm B (Placebo Comparator): Placebo (normal saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — 400mg Q2W intravenously
  Other Names: Anti epidermal growth factor receptor antibody h-R3
  Arms: Arm A
Drug: Placebo — Normal saline
  Other Names: Normal saline
  Arms: Arm B

SUMMARY:
There have been reports suggesting that anti-epidermal growth factor antibody nimotuzumab is advantageous for advanced esophageal cancer patients in combination with chemotherapy or radiotherapy. However, whether maintenance therapy of nimotuzumab provides benefit to advanced esophageal cancer patients is not known.

DETAILED DESCRIPTION:
We design this clinical trial to confirm the efficacy of maintenance treatment of nimotuzumab after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who was confirmed stage IV esophageal carcinoma by pathologic histology or cytology.
* The sample size estimate: 20 cases per arm.
* Males or females aged ≥18 years, < 75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Life expectancy ≥12 weeks.
* Males and females should be contraceptive during the period of the trial until 8 weeks after the last administration of the drug.
* Adequate bone marrow, renal, and liver function are required.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Institutional review board-approved informed consent will be obtained for every patient before initiation of any trial-specific procedure or treatment.

Exclusion Criteria:

* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Allergy to anti-EGFR antibody.
* Female subjects should not be pregnant or breast-feeding.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, or ≥ 50 ml/min. Adequate liver function: total bilirubin < 1.5 x upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PFS (Progression free survival) | 12 months

SECONDARY OUTCOMES:
Objective Response Rate | 6 months
Overall survival (OS) | 12 months
Disease control rate (DCR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, PhD, Principal Investigator — First Affiliated Hospital,Zhejiang University
Locations (2):
- China (2):
  - Qiong Zhao, Hangzhou, Zhejiang
  - The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang